CLINICAL TRIAL: NCT00275925
Title: A 24-Week Prospective, Open-Label, Multicenter Study to Evaluate the Effect on Seizure Frequency, Safety and Tolerability of Oxcarbazepine Monotherapy in Adult Patients With Partial Seizures
Brief Title: Safety and Efficacy of Oxcarbazepine Monotherapy in Adults With Partial Seizures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTRI476BRU01
Record Dates: First submitted 2006-01-11; First posted 2006-01-12 (Estimated); Last update posted 2007-11-30 (Estimated); Status verified 2007-11

CONDITIONS: Epilepsy, Partial Seizures
Keywords: partial epilepsy, oxcarbazepine, adults
MeSH Terms: conditions — Epilepsy; Seizures; Epilepsies, Partial | interventions — Oxcarbazepine

INTERVENTIONS:
Drug: Oxcarbazepine

SUMMARY:
This study is aimed to evaluate the efficacy, safety and tolerability of oxcarbazepine monotherapy in adults with partial seizures.

ELIGIBILITY:
Inclusion Criteria:

* males and females, 18 - 70 years of age;
* diagnosis of epilepsy, partial seizures;
* ineffective or intolerable present therapy with 1 antiepileptic drug, or none of previous therapy with antiepileptic drugs

Exclusion Criteria:

* progressive lesion of brain revealed by CT/MRI that performed no earlier than 2 years prior to screening;
* non-epileptic seizures;
* drug or alcohol dependence during a year prior to screening;

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2005-12; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Epileptic activity at electroencephalography in rest
Flash light and hyperventilation test with electroencephalography
Frequency of epileptic episodes according to patient's diary
Electrocardiogram analysis for rhythm and conduction
Blood test for sodium, hepatic enzymes and blood cells

SECONDARY OUTCOMES:
Quality of Life assessment at baseline, last visit
Tolerability and safety of 24 week's treatment with oxcarbazepine monotherapy in adult patients with partial seizures
Rate of patients with total and partial control of epilepsy
Rate of patients requiring additional antiepileptic drugs

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (7):
- Russia (7):
  - Epilepsy Department of the Moscow Research Institute of Psychiatry, Moscow
  - Neurology and Neurosurgery Department of the Moscow State Medico-stomatology University, Moscow
  - Neurology and Neurosurgery Department of the Russian State Medical University, Moscow
  - Neurology Department of I.M. Sechenov Moscow Medical Academy, Moscow
  - Neurology Department of Pediatric faculty of the Russian State Medical University, Moscow
  - Neurology Department of the Moscow region Research Institute named after M.F. Vladimirskiy, Moscow
  - Epilepsy Department of the V.M. Bekhterev Sant-Petersburg Psychoneurology Institute, Saint Petersburg